CLINICAL TRIAL: NCT06524570
Title: Treatment of Cancer with Immune Checkpoint Inhibition Therapy Boosted by High Intensity Focused Ultrasound Histotripsy; the IFOCUS Study
Brief Title: Treatment of Cancer with Immune Checkpoint Inhibition Therapy Boosted by High Intensity Focused Ultrasound Histotripsy
Acronym: iFOCUS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, K.P.M. Suijkerbuijk, Principal investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL85300.041.23
Record Dates: First submitted 2024-07-08; First posted 2024-07-29 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Metastatic Cancer
Keywords: Metastasized; Unresectable; Progressive after regular treatment
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Single arm phase 1 trial, monocenter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): High-intensity focused ultrasound histotripsy combined with ipilimumab + nivolumab
  Interventions: Device: HIFU-HT; Drug: ICI

INTERVENTIONS:
Device: HIFU-HT — High-Intensify Focused Ultrasound Histotripsy
Drug: ICI — Ipilimumab and nivolumab
  Other Names: Immune checkpoint inhibitors

SUMMARY:
This phase 1 clinical trial aims to evaluate the safety, tolerability and feasibility of combination treatment of High Intensity Focused Ultrasound Histotripsy (HIFU-HT) and immune checkpoint inhibitors (ICI) in adult patients with metastatic or unresectable cancer that have progressive disease after regular treatment. Patients will undergo one single session of HIFU-HT during treatment with ipilimumab and nivolumab. Safety, tolerability and feasibility endpoints will be studied as well as radiologic, immunologic and clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic or unresectable cancer that progressed under standard of care treatment options.
2. Age ≥ 18 years.
3. Has signed and dated written informed consent before performing any study procedure, including screening.
4. Anticipated life expectancy ≥ 12 weeks by investigator judgement.
5. At least one tumor lesion (primary tumor or metastasis) which is amenable to application of high intensity focused ultrasound histotripsy (determined by a radiologist with HIFU-expertise).

   * The lesion must have a distance of ≤30 mm to the skin.
   * At least part of the lesion must have a distance of ≥10 mm to the skin and other vulnerable structures (e.g. large blood vessels). This part should be sufficient to be able to select at least one HT focus in an area of solid tumor.
   * If the target lesion contains cystic or necrotic regions: the solid component should be ≥10 mm in diameter, sufficient to be able to select at least one HIFU-HT focus in an area of solid tumor with ≥10 mm distance to the skin.
6. Sonication will be performed on tumors that have not previously directly been treated with radiation therapy or surgery unless they showed significant mass regrowth.
7. Measurable disease (at least one lesion besides the HIFU-HT treated lesion) on CT according to RECIST V 1.1 criteria (or on PET-CT according to PERCIST criteria) as assessed by investigator and local radiology review.
8. Performance status of 0 or 1 on the WHO Performance Scale.
9. Screening laboratory values must meet the following criteria:

   * WBC ≥ 2.0x109/L,
   * Neutrophils ≥1.5x109/L
   * Platelets ≥100 x109/L
   * Hemoglobin ≥5.5 mmol/L
   * Serum creatinine ≤1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥60 mL/minute (≤Grade 1)
   * Aspartate aminotransferase (AST) ≤2.5 x ULN; alanine aminotransferase (ALT) ≤2.5 x ULN; AST/ALT <5 x ULN if liver involvement
   * Serum bilirubin ≤1.5 x ULN or direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5xULN, except in subjects with Gilbert's Syndrome
10. Patients must agree to use an adequate method of contraception for the course of the study through 180 days after the last dose of study medication.
11. Patients must be willing to undergo tumor biopsy.

Exclusion Criteria:

1. Presence of known central nervous system, meningeal, or epidural metastatic disease. However, subjects with known brain metastases are allowed if the brain metastases are stable for ≥4 weeks before the first dose of study treatment. Stable is defined as neurological symptoms not present or resolved to baseline, no radiologic evidence of progression, and steroid requirement of prednisone ≤10 mg/day or equivalent.
2. Patients currently participating and receiving study therapy or patients who participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of the study treatment.
3. Prior chemotherapy, targeted small molecule therapy or monoclonal antibodies within 4 weeks prior to the first dose of the study treatment.
4. Prior radiotherapy within 8 weeks prior to the first dose of the study treatment. The patient will be excluded from the study if the only targetable lesion has directly been treated with radiation therapy in the past with an exception for lesions that showed massive regrowth.
5. Prior surgery or ablative therapy within 4 weeks prior to the first dose of the study treatment. The patient will be excluded from the study if the only targetable lesion has directly been treated with ablative therapy in the past.
6. Ongoing adverse events > Grade 1 due to a previously administered therapy. Subjects with ≤ Grade 2 neuropathy, vitiligo, thyroid disorders, hypocortisolism or alopecia of any grade are an exception to this criterion and may qualify for the study.
7. History of other malignancies, except adequately treated and a cancer-related life-expectancy of more than 5 years.
8. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids; exceeding prednisolone 10 mg or equivalent.
9. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, high-dose corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Active infection requiring systemic therapy.
11. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
12. Known history of active Tuberculosis.
13. Receipt of a live vaccine within 4 weeks prior to the first dose of the study treatment.
14. Hypersensitivity to any of the study drugs or their excipients.
15. Contra-indications to MR imaging (e.g. certain pacemakers or severe claustrophobia). Contra-indications to gadolinium-based contrast agents are not an exclusion criterion, as a different brand of gadolinium can be used or if necessary the MRI can be performed without contrast.
16. Pregnancy or lactation.
17. Any other medical or social condition that, in the opinion of the Principal Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Number and severity of adverse events until 100 days after the last study treatment | Adverse events will be assessed up to 100 days after the last study treatment
  Safety: Incidence and severity of adverse events (related to HIFU-HT or the combination of HIFU-HT and ICI.)
Tolerability: Discontinuation rate | At every visit untill 2 years after first study treatment
  Discontinuation rate due to adverse events.
Tolerability: Patient reported tolerability by HIFU-HT-tolerability questionnaire | Day 8 + 15
  The HIFU-HT tolerability questionnaire is a self-reported, customized questionnaire that describes the burden/complaints a respondent experienced following HIFU-histotripsy treatment. The questionnaire comprises questions about pain, use of pain medication, complaints other than pain, burden of MRI scan, burden of peri-procedural analgesia, time burden of treatment. Respondents are asked to grade the experienced complaints or burden on a scale of 5 options, ranging from no complaints/no burden to severe complaints/severe burden. If respondents report pain, they are asked to grade their pain on a scale ranging from 0 - 10 (0 reflecting no pain, 10 reflecting worst possible pain) and respondents are asked for how many days the pain was present (ranging from 0 to 7 days).
Tolerability: Patient reported tolerability by EQ-5D | Baseline, days 1, 8, 15, 22, 43, 64, 91; thereafter every 4 to 8 weeks until 2 years after start of therapy
  The EuroQol Group EQ-5D questionnaire (Dutch version) is a self-reported questionnaire that reflects a respondent's health. The EQ-5D comprises questions on 5 domains (mobility, self care, daily activities, pain/complaints, mood), for each of these domains respondents state whether they have no problems, some problems or severe problems. Respondents are also asked to grade their general health status on a scale of 0 - 100 (0 reflecting the worst possible health status, 100 reflecting the best possible health status).
Tolerability: Patient reported tolerability by USD-I | Baseline, days 1, 8, 15, 22, 43, 64, 91; thereafter every 4 weeks until 2 years after start of therapy
  The Utrecht symptom diary immunotherapy (USD-I) is a self-reported questionnaire that was developed and validated in the UMC Utrecht to score symptoms patients might experience during/after treatment with checkpoint inhibition therapy. The questionnaire comprises of questions on 19 possible symptoms (apetite, stool pattern, diarrhea, abdominal pain, coughing, eye complaints, skin rash, pruritus, headache, myalgia, arthralgia, paresthesias, pain, sleeping problems). Respondents are asked to grade these symptoms on a scale of 0 - 10 (0 reflecting no problems, 10 reflecting worst possible problem).
Feasibility: Number of technically effective HIFU-HT procedures | Day 8
  Feasibility: The number of technically effective HIFU-HT procedures.
Feasibility: Percentage of screening failures | Baseline
  Feasibility:The percentage screening failures.
Feasibility: Time burden | Through study completion, up to two years after start of study treatment
  Feasibility: Time burden of the study procedures.

SECONDARY OUTCOMES:
Radiological response: MRI | Directly after HIFU-HT and 12 weeks after start of treatment
  Local response of HIFU-HT treated tumor as assessed by MRI directly and 12 weeks after HIFU-HT
Radiological response: CT | 12 weeks after start of treatment; every 12 weeks while on treatment up to two years after start therapy
  Best overall systemic response using RECIST 1.1 as assessed by CT-scan every 12 weeks (or using PERCIST as assessed by PET-CT if not RECIST measurable)
Immunologic response | Baseline and days 1, 8, 9, 15, 22, 64
  1. Analysis of immunological parameters in peripheral blood
  2. Analysis of immune infiltrates in tumor biopsies taken at baseline and 7 days after HIFU-HT
Overall survival | Every 12 weeks until 2 years
  Explorative analysis to assess overall survival in months while taking into consideration the heterogeneous patient population in this basket design.
Progression free survival | Every 12 weeks until 2 years
  Explorative analysis to assess progression-free survival in months while taking into consideration the heterogeneous patient population in this basket design.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No